CLINICAL TRIAL: NCT05480176
Title: The National Chronic Obstructive Pulmonary Disease Screening Program in China
Brief Title: The China National COPD Screening Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof., China-Japan Friendship Hospital
Other Study IDs: 2021-145-K103
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Screening; Spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-COPD high-risk population: The local residents gain a COPD-SQ score < 16.
  Interventions: Other: Comprehensive intervention and management Ⅰ
- COPD high-risk population: The participants have a COPD-SQ score ≥ 16 with a FEV1/FVC ≥ 0.70 either with or without bronchodilator administration.
  Interventions: Other: Comprehensive intervention and management Ⅱ
- Confirmed COPD patients: The participants have a COPD-SQ score ≥ 16 with a FEV1/FVC ≥ 0.70 after administration of bronchodilators.
  Interventions: Other: Comprehensive intervention and management Ⅲ

INTERVENTIONS:
Other: Comprehensive intervention and management Ⅰ — Mainly health advisory.
  Groups: Non-COPD high-risk population
Other: Comprehensive intervention and management Ⅱ — Health advisory and regular follow-ups.
  Groups: COPD high-risk population
Other: Comprehensive intervention and management Ⅲ — Pharmaceutical and non-pharmaceutical (e.g. health advisory, rehabilitation, etc.) interventions according to standardized clinical guidelines, with regular follow-ups.
  Groups: Confirmed COPD patients

SUMMARY:
The national COPD screening program is in a cross-sectional manner at the baseline, planning to recruit a total of 800,000 participants from 160 districts or counties (5,000 for each site on average) from 31 provinces, autonomous regions or municipalities directly under the central government of China. The filtered COPD high-risk population and confirmed COPD patients will be managed and followed up according to the standardized clinical guidelines. The major aims of the program are to estimate the prevalences of COPD high-risk population and under- or miss- diagnosed COPD patients, and to manage the development and outcomes of the disease.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 35 and 75 years;
* residents living in the survey area with more than 6 months in the past year.

Exclusion Criteria:

* experienced myocardial infarction, stroke or shock in the past 3 months;
* experienced severe cardiac insufficiency, severe arrhythmia or unstable angina pectoris in the past 4 weeks;
* experienced massive hemoptysis in the past 4 weeks;
* received chest, abdominal or ophthalmic surgery in the past 3 months;
* have mental disorders (e.g. auditory hallucinations, visual hallucinations, taking antipsychotics, seizures requiring medication, etc.);
* have cognitive impairment (e.g. dementia, comprehension impairment, etc.);
* have uncontrolled hypertension (i.e. systolic blood pressure > 200 mmHg, diastolic blood pressure > 100 mmHg);
* present with heart rate >120 beats/min;
* have aortic aneurysm;
* have severe hyperthyroidism;
* are pregnant or lactating women;
* experienced respiratory infectious diseases (e.g. tuberculosis, influenza, etc.) in the past month.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are potentially under a high risk of suffering COPD with an age between 35 and 75 years are eligible to be recruited. The participants should be residents who were living in the survey area with more than six months in the past year.
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung function | 2 years
  The changes of lung function (e.g. FEV1, FVC, FEV1/FVC, etc.) (P.S.: it is hard to assume that the lung function would be improved or decling, especially for the pre- or early-COPD population)

SECONDARY OUTCOMES:
Respiratory symptoms | 2 years
  The appearance frequencies of respiratory symptoms (e.g. cough, sputum, wheeze, dyspnea, etc.)
Exacerbations | 2 years
  The numbers of exacerbations (e.g. emergency department visit, hospital admission, etc.) that related to COPD

CONTACTS AND LOCATIONS:
Overall Officials: Ting YANG, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data would be available on reasonable request from the principal investigator.